CLINICAL TRIAL: NCT02772913
Title: Acute Mesenteric Ischemia in the Emergency Department: Incidence, Early Recognition and Risk Stratification From an Observational Multicenter Study
Brief Title: Mesenteric Ischemia in the Emergency Department: a Retrospective Multicenter Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Genova (Other)
Collaborators: University of Bari (Other); University of Siena (Other)
Responsible Party: Principal Investigator, Stefano Sartini, Medical doctor, Consultant in Emergency Medicine, University of Genova
Other Study IDs: RetroMesIsch
Record Dates: First submitted 2016-03-24; First posted 2016-05-16 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Acute Mesenteric Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- acute mesenteric ischemia: patients with abdominal pain and acute mesenteric ischemia
- non-acute mesenteric ischemia: patients with abdominal pain without mesenteric ischemia

SUMMARY:
Acute mesenteric ischemia is a life-threatening condition characterized by high mortality if unrecognized early. This multicenter retrospective observational study will review the emergency departments's (ED) notes of all patients discharged from hospital with a diagnosis of acute mesenteric ischemia in 2014-2015 comparing it with those admitted to the ED for abdominal pain in the same timeframe.

DETAILED DESCRIPTION:
Acute mesenteric ischemia is a condition characterized by non-specific presentation (typical clinical presentation is considered "abdominal pain out of proportion to examination") that may be under-recognized in the Emergency Department. Early identification and treatment is essential to improve outcome as mortality rate is attested around 80% if untreated within few hours from onset. The investigators aim to review the emergency department's clinical notes of patients discharged from hospital in 2014 and 2015 diagnosed with acute mesenteric ischemia. Furthermore the investigators will consider patients admitted for "abdominal pain" in the same time frame without acute mesenteric ischemia and we will compare presentation symptoms, medical history, medications, vitals, laboratory markers and imaging finding of the two groups. From this comparison, the investigators will be able to clarify the incidence among general population and among patients presenting acute abdominal pain. Finally, using multivariate analysis, the investigators may identify those variables predictive of acute mesenteric ischemia. This study will be held in three university hospitals and all data analyzed together.

ELIGIBILITY:
Inclusion Criteria:

* ICD-9 diagnosis of acute mesenteric ischemia in 2014 and 2015
* Admitted to hospital after Emergency Department assessment
* age>18

Exclusion Criteria:

* age<18
* post-traumatic or post-surgery related acute mesenteric ischemia
* lack of assessment in the Emergency Department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients discharged from hospital with ICD-9 code related to acute mesenteric ischemia (1st cohort) compared with patients admitted for acute abdominal pain
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-06 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | 30 days from hospital admission

SECONDARY OUTCOMES:
in-hospital adverse outcome: cardiac arrest, ICU admission, septic shock, major bleeding. | 30 days from hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Savarino, Professor, Study Chair — University of Genova
Locations (1):
- IRCCS San Martino, Genoa, Liguria, Italy

IPD SHARING:
Plan to Share IPD: Yes